CLINICAL TRIAL: NCT03522415
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of HLX01 (Recombinant Human-mouse Chimeric Anti-CD20 Monoclonal Antibody Injection) Combined With MTX Therapy in Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate
Brief Title: Study of Safety and Efficacy of HLX01+MTX in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX01-RA03
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Moderately to Severely Active Rheumatoid Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX01+MTX (Experimental)
  Interventions: Drug: HLX01; Drug: Methotrexate（MTX）
- Placebo+MTX (Placebo Comparator)
  Interventions: Drug: Methotrexate（MTX）

INTERVENTIONS:
Drug: HLX01 — HLX01,Recombinant Human-mouse Chimeric Anti-CD20 Monoclonal Antibody Injection is recombinant human-mouse chimeric anti-cd20 CD20 monoclonal antibody.
  Arms: HLX01+MTX
Drug: Methotrexate（MTX） — Methotrexate is a slow-acting antirheumatic drug.

SUMMARY:
To compare the efficacy between the HLX01 group and the placebo group through the proportion of subjects meeting the ACR20 improvement criteria for remission

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are voluntary to participate in the study and sign a written ICF, and willing and able to follow the study protocol (e.g. able to understand and complete the questionnaire, follow the visit plan and use the drug).
2. 18 years ≤ age ≤75 years, male or female.
3. Subjects who are diagnosed with moderately to severely active RA with a course of disease of at least 6 months, DAS28 CRP > 3.2 at Screening, and at least 6 swollen joints (based on 66 joints) and 6 tender joints (based on 68 joints) at Screening and Baseline (Day 1) visit. If a joint has both swollen and tender symptoms, then this joint should be included in both the SJC and TJC (except for artificial joints).
4. MTX-IR: Subjects must be currently receiving MTX 10-25 mg/week for at least 12 weeks and have been on a stable dose for at least 4 weeks prior to study entry (Day 1). MTX needs to be given at a stable dose throughout the study, unless dose adjustments are made for safety reasons.
5. The accepted RA treatment must meet the following conditions:

   1. Subjects are willing to receive oral folic acid therapy (at least 5 mg/week or at a dose determined based on local medical practice) or equivalent medications (combination medications necessary for MTX therapy) during the entire study, and the dose of folic acid or equivalent medications should be stable for a minimum of 4 weeks prior to the start of study treatment (Day 1).
   2. If the subject has been previously treated with traditional disease-modifying anti-rheumatic drugs (DMARDs) other than MTX: leflunomide should be discontinued at least 8 weeks prior to the start of study treatment (Day 1), but if they have received standard cholestyramine elution treatment for 11 days, leflunomide will need to be discontinued at least 4 weeks prior to the start of study treatment (Day 1); other DMARDs will need to be discontinued at least 4 weeks prior to the start of study treatment (Day 1). These drugs are not allowed to be used throughout the study.

      * Standard cholestyramine elution treatment: cholestyramine 8 g orally, three times daily for 11 consecutive days.
   3. If the subject is being treated with Tripterygium wilfordii, the drug should be discontinued at least 2 weeks prior to the start of study treatment (Day 1) and is not allowed to be used throughout the study.
   4. If the subject is receiving oral glucocorticoid treatment, the dose should not exceed prednisolone 10 mg/day (or equivalent dose of other glucocorticoids), and the dose should have been stable for at least 4 weeks prior to the start of study treatment (Day 1) and remain stable throughout the 24-week treatment period (except for those receiving rescue treatment); if already discontinued, oral glucocorticoids should have been discontinued for at least 2 weeks prior to the start of study treatment (Day 1).
   5. Glucocorticoid treatment via intra-articular or injection administration is not allowed within 6 weeks prior to the start of study treatment (Day 1) and during treatment (until Week 24), except for methylprednisolone 80 mg intravenously administered prior to study drug infusion (as this is part of the study process).
   6. Any non-steroidal anti-inflammatory drugs (NSAIDs) must have been on a stable dose for a minimum of 2 weeks prior to the start of study treatment (Day 1) and remain on a stable dose throughout the 24-week treatment period (except for those receiving rescue treatment); if already discontinued, NSAIDs should have been discontinued for at least 2 weeks prior to the start of study treatment (Day 1).
6. Eligible subjects must meet the following screening criteria for tuberculosis:

   1. The subject has no active tuberculosis.
   2. The subject has no occult tuberculosis infection.
   3. QUANTIFERON®-TB Gold test is negative at Screening.
   4. If the QUANTIFERON®-TB Gold test result is indeterminate, a repeat test is needed. If it is still indeterminate upon retest, the Investigator should make a comprehensive judgment based on the subject's symptoms and signs, history of exposure to TB patients and chest X-ray examination. If active tuberculosis is excluded, the subject can be enrolled.
7. Women of childbearing potential * must agree to take reliable contraceptives during the study and 12 months following trial completion or termination (e.g., hormonal contraception pills, contraceptive patches, IUDs, physical contraception). (Note: * Subjects without childbearing potential refer to female subjects who have been menopausal for at least 2 years or have undergone total hysterectomy, bilateral tubal ligation or bilateral salpingo-tubal resection and/or bilateral ovariectomy, or who have congenital infertility.)
8. Men whose partners are women of childbearing potential are required to take reliable contraception during th study and 12 months following trial completion or termination, and the male subject will not donate sperm.

Exclusion Criteria:

1. Previously used TNF-α antagonists, other biologics for RA, or targeted synthesized DMARDs (e.g., JAKs enzyme inhibitor tofacitinib).
2. ACR functional Class IV or bedridden/wheelchair-bound for a long term.
3. Primary or secondary immunodeficiency in previous or current medical history, including know history of HIV infection and positive HIV.
4. Moderate to severe congestive heart failure (Class III or IV of New York Heart Association ).
5. Interstitial lung disease (except mild).
6. Known allergic to murine proteins or other antibodies.
7. History of malignancy, including solid tumors, hematologic tumors and carcinoma in situ(except subjects with previous resected and cured basal or cutaneous squamous cell carcinoma, cervical dysplasia or in situ grade I cervical cancer at least 12 months prior to the Screening Visit).
8. Receipt a live vaccine/attenuated vaccine within 12 weeks prior to the Screening Visit until Week 48.
9. Any disease or treatments (including biotherapy) that, at the discretion of the Investigator, may bring unacceptable risk to the subject.
10. Pregnant or nursing female subjects, or subjects will pregnant or breastfeeding during the study period or within 12 months of the last dose.
11. Previously or currently suffering from inflammatory joint diseases other than RA (e.g. gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathies, Lyme disease, etc.), or other systemic autoimmune diseases (e.g., systemic lupus erythematosus, inflammatory bowel disease, pulmonary fibrosis, Felty's syndrome, scleroderma, inflammatory myopathy, mixed connective tissue disease, or any overlap syndromes).
12. Evidence significant unconcomitant diseases, such as, but not limited to, nervous system, cardiovascular, renal, hepatic, endocrine or gastrointestinal diseases which would preclude patient participation at the discretion of the Investigator.
13. Positive anti-Hepatitis C virus (HCV) antibody at Screening.
14. Positive anti-Treponema pallidum (TP) antibody at Screening.
15. Positive hepatitis B surface antigen (HBsAg) at the Screening; a subject negative for HBsAg yet positive for hepatitis B core antibody (HBcAb) must be further tested for hepatitis B virus (HBV) deoxyribonucleic acid (DNA); only HBV DNA-negative subjects can be enrolled.
16. Any active infection (except nail bed fungal infection), or any serious infection requiring hospitalization or intravenous anti-infection treatment within 4 weeks before the screening visit; or oral anti-infective drug treatment within 2 weeks before the screening visit.
17. History of deep gap/tissue infections (e.g., fasciitis, abscess, osteomyelitis) within 52 weeks prior to the screening visit.
18. History of serious or opportunistic infections in the recent two years at the discretion of the Investigator.
19. History of chronic infections (e.g., chronic pyelonephritis, bronchiectasis or osteomyelitis).
20. Any congenital or acquired neurological, vascular or systemic disease that may affect any of the efficacy evaluations in this study, especially joint pain and swelling (e.g., Parkinson's disease, cerebral palsy, diabetic neuropathy).
21. History of alcohol or drug abuse within 52 weeks prior to the Screening Visit or subjects currently with alcohol or drug abuse (at the discretion of the Investigator).
22. Received anti-integrin αV antibody or cell depletion therapy including B-cell depletion therapy(e.g., CD20+, or CD19+, or CD38+ cell depletion) within 3 months or 5 half-lives(whichever is longer) prior to the screening visit.
23. Intolerant of glucocorticoid injections or have contraindications to glucocorticoids.
24. Have any of the following specific abnormalities on screening laboratory tests:

    1. Aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN);
    2. Alanine aminotransferase (ALT)> 2 × ULN;
    3. Hemoglobin <8.0 g/dL;
    4. Absolute neutrophil count <1.5 × 109/L;
    5. Platelet count <75 × 109/L;
    6. White blood cell count <3 × 109/L;
    7. Serum creatinine> 1.5 × ULN. * No medical supportive treatments (e.g. various WBC-increasing drugs, anemia drugs (except folic acid), hepatoprotective and enzyme-lowering drugs, blood transfusions, etc.) are allowed within 2 weeks prior to screening.
25. Participated in any clinical study (within 12 weeks or with the 5 half-lives of the study drug, whichever is longer) before the screening visit, or subjects planning to participate in other clinical studies during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
ACR20 | 24 weeks
  Proportion of subjects meeting the ACR20

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Jiujiang No.1 peoples's hospital, Jiujiang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zeng X, Liu J, Liu X, Wu L, Liu Y, Liao X, Liu H, Hu J, Lu X, Chen L, Xu J, Jiang Z, Lu FA, Wu H, Li Y, Wang Q, Zhu J; HLX01-RA03 Investigators. Efficacy and safety of HLX01 in patients with moderate-to-severe rheumatoid arthritis despite methotrexate therapy: a phase 3 study. Arthritis Res Ther. 2022 Jun 10;24(1):136. doi: 10.1186/s13075-022-02821-x. PMID 35689239
- See also: Annals of the Rheumatic Diseases 2021;80:1122-1123. — http://dx.doi.org/10.1136/annrheumdis-2021-eular.282